CLINICAL TRIAL: NCT03549858
Title: Patient Reported Outcomes Burdens and Experiences (PROBE) - Phase 3 - Longitudinal Data Collection
Brief Title: Patient Reported Outcomes Burdens and Experiences - Phase 3
Acronym: PROBE-3
Status: Recruiting | Type: Observational
Sponsor: McMaster University (Other)
Collaborators: Patient Outcomes Research Group (PORG) (Unknown); National Hemophilia Foundation (Unknown)
Responsible Party: Sponsor
Other Study IDs: PROBE-3
Record Dates: First submitted 2018-05-15; First posted 2018-06-08 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Hemophilia; Chronic Disease
MeSH Terms: conditions — Hemophilia A; Chronic Disease | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Quality of life measure (survey) — The QoL tool is a questionnaire

SUMMARY:
The PROBE Phase-3 study will collect data on patient reported outcomes, burdens, and experiences in patients living with hemophilia. The investigators will perform comparisons among countries, within country over time, within country against national normative data.

DETAILED DESCRIPTION:
BACKGROUND

The PROBE questionnaire is a tool for the assessment of patient-reported outcome, burdens and experiences. Until now, it has been used in persons living with hemophilia (PWH) and healthy controls. In phase 1 of the study, the investigators developed the questionnaire. In phase 2 of the study, the investigators evaluated the reliability, reproducibility, responsiveness, and costs of PROBE. The tool has been tested across 21 countries and it has been shown that PROBE is a valid questionnaire for the evaluation of patient reported outcomes (PROs) in PWH and control populations. The questionnaire is available in 11 languages (with 20 localized versions worldwide), and another 17 languages and 45 more localizations are in the process of development.

CURRENT STUDY and FUTURE DIRECTIONS

Phase 3 is the natural prosecution of the project. In this phase, the investigators aim at maintaining the capacity to collect data on PROBE, and the infrastructure will also be modified in order to allow for longitudinal collection of PROBE data (in previous phases, the investigators only collected anonymized data).

The objective of the study is to compare data on PROBE between countries, within-countries over time, and within-countries against national normative data. Reports will be produced every 2 years. Data collected during phase 2 of the study will also be used.

At the same time, the research framework will have the potential for:

* Expanding country participation within existing and new regions.
* Integrating the PROBE questionnaire in clinical trials, longitudinal studies, health technology assessment studies, routine clinical care, and registries.
* Using PROBE in new countries
* Testing the performance of the PROBE questionnaire in new patient populations

INVESTIGATION TEAM

Principal Investigator:

1. Mark Skinner JD, Institute for Policy Advancement Ltd. (US)

   Co-Investigators:
2. Alfonso Iorio MD Ph.D. FRCPC, McMaster University, Department of Clinical Epidemiology and Biostatistics (Canada)
3. Randall Curtis MBA, Factor VIII Computing (US)
4. Neil Frick MS, National Hemophilia Foundation (US)
5. Michael Nichol Ph.D., University of Southern California, School of Policy and Planning Development (US)
6. Declan Noone, Irish Hemophilia Society (Ireland)
7. David Page, Canadian Hemophilia Society (Canada)
8. Jeff Stonebraker Ph.D., North Carolina State University Poole College of Management (US)
9. Brian O'Mahoney, Irish Hemophilia Society (Ireland)
10. Chatree Chai-Adisaksopha, MD MSc.

ELIGIBILITY:
Inclusion Criteria:

* PWH will be recruited through national hemophilia patient organizations utilizing their existing membership rosters, social media outlets and meetings / events. The investigators are not proposing a pre-determined method of PWH recruitment. They will utilize the information acquired in the workshop and take-home project to inform best practice in recruitment methodology for the study. The investigators may consider requesting different countries test different PWH recruitment strategies to test reproducibility.

In the future, the questionnaire might also be administered to patients with other chronic conditions.

Exclusion Criteria:

* Disease severity and Age bands or age limits (e.g. ≥ Age 18) may be utilized to narrow the study population.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Moderate / Severe PWH (Age bands or limits may be utilized to narrow the study population). Patients will be recruited according to the final inclusion criteria. No randomization will be required. Two moderate to large test runs of the inventory will be conducted in each country three months apart to demonstrate reproducibility. PWH participating in each of the two test runs may, but would not necessarily be the same.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Between-countries variability of the PROBE score | 2 years
  Mean difference and standard deviation of the PROBE score between countries.

SECONDARY OUTCOMES:
Within-countries variability of the PROBE score | 2 years
  Mean difference and standard deviation of the PROBE score in repeated assessments within countries.
Within-countries comparison of the PROBE score in PWH against national normative data | 2 years
  Mean difference and standard deviation of the PROBE score in PWH against national normative data within countries.

CONTACTS AND LOCATIONS:
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

REFERENCES:
- [Background] Skinner MW, Chai-Adisaksopha C, Curtis R, Frick N, Nichol M, Noone D, O'Mahony B, Page D, Stonebraker JS, Iorio A. The Patient Reported Outcomes, Burdens and Experiences (PROBE) Project: development and evaluation of a questionnaire assessing patient reported outcomes in people with haemophilia. Pilot Feasibility Stud. 2018 Feb 27;4:58. doi: 10.1186/s40814-018-0253-0. eCollection 2018. PMID 29497561